CLINICAL TRIAL: NCT05718193
Title: Real-Time Artificial Intelligence Assissted Colonoscopy to Identify and Classify Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Loudi Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 202112254
Record Dates: First submitted 2023-01-03; First posted 2023-02-08 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-01

CONDITIONS: Artificial Intelligence; Colonoscopy; Quality Control

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The DeFrame Group (Experimental): Subjects in the DeFrame group were treated with a real-time computer-aided polyp detection system named DeFrame during colonoscopy.
  Interventions: Diagnostic Test: DeFrame
- The Classified DeFrame Group (Experimental): Subjects in the Classified DeFrame group were treated with a real-time computer-aided polyp detection and classification system named Classified DeFrame during colonoscopy.
  Interventions: Diagnostic Test: Classified DeFrame
- The Control Group (Experimental): Subjects in the control group underwent standard colonoscopy.
  Interventions: Diagnostic Test: conventional colonoscopy

INTERVENTIONS:
Diagnostic Test: DeFrame — The DeFrame system is applicated during colonoscopy. The DeFrame system superimposes a rectangular box on the polyp lesion area in the colonoscopy field of view, notifying the endoscopists of the presence of the lesion.
  Arms: The DeFrame Group
Diagnostic Test: Classified DeFrame — The Classified DeFrame system is applicated during colonoscopy. The Classified DeFrame system superimposes a rectangular box on the polyp lesion area in the colonoscopy field of view, the color of the rectangle box will turn blue when the polyp is considered as an adenoma, notifying the endoscopists of the presence of the lesion.
  Arms: The Classified DeFrame Group
Diagnostic Test: conventional colonoscopy — conventional colonoscopy
  Arms: The Control Group

SUMMARY:
To investigate the degree of the real-time detection and classification system for increasing the adenoma detection rate during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 to 85 years old. Colonoscopies for primary CRC screening of the subjects are required.

Exclusion Criteria:

History of CRC,inflammatory bowel disease, previous colonic resection, antithrombotic therapy precluding polyp resection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2868 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate | up to 9 months
  Percentage of patients who have 1 or more histologically confirmed adenoma resected divided by the total number of colonoscopies.
adenomas per colonoscopy | up to 9 months
  Total number of histologically confirmed adenomas resected divided by the total number of colonoscopies.

CONTACTS AND LOCATIONS:
Overall Officials: xiaowei liu, doctor, Study Director — Xiangya Hospital of Central South University
Locations (2):
- China (2):
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Loudi Central Hospital, Loudi, Hunan

IPD SHARING:
Plan to Share IPD: No